CLINICAL TRIAL: NCT06880861
Title: Investigating Memory and Physical Activity After Cancer Treatment in Survivors of Adolescent and Young Adult Cancers
Acronym: IMPACT
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-008654; NCI-2025-01193 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-008654 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
Keywords: cancer; adolescent; young adult; cognition; memory; exercise; physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete questionnaires and cognitive tasks and wear an activity monitor to measure physical activity on study. Some patients may optionally participate in an interview on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates relationships among physical activity, thinking, and memory after cancer treatment in survivors of adolescent and young adult cancers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18+ years)
* Primary diagnosis of cancer when 15-39 years-old
* Access to a desktop computer or laptop with reliable internet access
* No gross motor impairments that prohibit ambulation
* Willing to complete study requirements
* English speaking

Exclusion Criteria:

* Diagnosed with nonmelanoma skin cancer only
* Not diagnosed with cancer in adolescent and young adult (AYA) age range of 15-39 years
* Scheduled travel during the study period that is not indicative of individual's normal schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary diagnosis of cancer when 15-39 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance on Stroop task | Up to 4 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games"). CNS Vital Signs is a computerized neuropsychological/neurocognitive assessment platform used by clinicians and researchers to objectively evaluate brain function and neurocognitive status, offering a range of tests and tools for assessment and management of various neurological and behavioral conditions.

SECONDARY OUTCOMES:
Cognitive performance on Visual Memory Test | 2 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games"). CNS Vital Signs is a computerized neuropsychological/neurocognitive assessment platform used by clinicians and researchers to objectively evaluate brain function and neurocognitive status, offering a range of tests and tools for assessment and management of various neurological and behavioral conditions.
Cognitive performance on Verbal Memory Test | 2 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games"). CNS Vital Signs is a computerized neuropsychological/neurocognitive assessment platform used by clinicians and researchers to objectively evaluate brain function and neurocognitive status, offering a range of tests and tools for assessment and management of various neurological and behavioral conditions.
Cognitive performance on Symbol Digit Coding Test | 2 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games"). CNS Vital Signs is a computerized neuropsychological/neurocognitive assessment platform used by clinicians and researchers to objectively evaluate brain function and neurocognitive status, offering a range of tests and tools for assessment and management of various neurological and behavioral conditions.
Cognitive performance on Shifting Attention Test | 2 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games"). CNS Vital Signs is a computerized neuropsychological/neurocognitive assessment platform used by clinicians and researchers to objectively evaluate brain function and neurocognitive status, offering a range of tests and tools for assessment and management of various neurological and behavioral conditions.
Cognitive performance on Continuous Performance Test | Up to 4 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games").
Cognitive performance on Reasoning Test | 2 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games"). CNS Vital Signs is a computerized neuropsychological/neurocognitive assessment platform used by clinicians and researchers to objectively evaluate brain function and neurocognitive status, offering a range of tests and tools for assessment and management of various neurological and behavioral conditions.
Cognitive performance on Four Part Continuous Performance Test | 2 weeks
  Assessed using the CNS Vital Signs computerized testing platform ("brain games"). CNS Vital Signs is a computerized neuropsychological/neurocognitive assessment platform used by clinicians and researchers to objectively evaluate brain function and neurocognitive status, offering a range of tests and tools for assessment and management of various neurological and behavioral conditions.
Self-reported cognition - FACT-COG | 2 weeks
  Evaluated using the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG), a 37-item questionnaire assessing cognitive impairment, cognitive abilities, and quality of life over the past 7 days. Responses are on a 5-point scale (Never; About once a week; Two to three times a week; Nearly every day; Several times a day). Higher scores generally indicate better self-reported cognition.
Average weekly minutes of physical activity | 2 weeks
  Moderate-to-vigorous physical activity (MVPA) will be measured using an accelerometer (activPAL) which participants will wear on their non-dominant thigh for 7 consecutive days.

CONTACTS AND LOCATIONS:
Overall Officials: Diane K. Ehlers, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, limited datasets will be shared with other researchers upon request or according to journal publication requirements
Supporting Information: Study Protocol
Time Frame: At time of first publication (as required by journals) until last manuscript is published.
Access Criteria: If required by journal and case by case upon request to the PI

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials